CLINICAL TRIAL: NCT05599646
Title: Effects of Gamified Versus Traditional Pedometer-Based Walking Intervention on Physical Activity, Fatigue and Sleep Quality Among Hemodialysis Patients: A Quasi-Experimental Study
Brief Title: Pedometer-Based Walking Intervention on Physical Activity Among Hemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, mohamed elsayed hamed elzeky, lecturer at medical surgical nursing, Mansoura University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: mans
Record Dates: First submitted 2022-10-24; First posted 2022-10-31 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2024-03

CONDITIONS: Physical Inactivity; Fatigue
MeSH Terms: conditions — Sedentary Behavior; Fatigue

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- traditional pedometer group (Experimental)
  Interventions: Behavioral: traditional pedometer based walking intervention
- gamified smartphone pedometer group (Experimental)
  Interventions: Behavioral: gamified pedometer based walking intervention
- control group (No Intervention)

INTERVENTIONS:
Behavioral: traditional pedometer based walking intervention — Participants were recommended to monitor their step count using traditional pedometer and to increase their steps by 10% compared with the prior week. the intervention will continue for 12 weeks
  Arms: traditional pedometer group
Behavioral: gamified pedometer based walking intervention — Participants were recommended to monitor their step count using gamified pedometer, earn money, compete friends and to increase their steps by 10% compared with the prior week. the intervention will continue for 12 weeks
  Arms: gamified smartphone pedometer group

SUMMARY:
Patients undergoing HD are mostly physically inactive and have reduced functional capacities compared to healthy individuals which contributes to a decreased quality of life and consequently increases the risk of mortality

DETAILED DESCRIPTION:
Physical activity has been shown to have various positive effects on HD patients . Some of the important benefits linked to exercise include an improvement in physical fitness , aerobic capacity , dialysis adequacy (measured as urea Kt/V) , quality of life , and reduced depressive symptoms .Walking can be considered as the most natural form of PA as it is easily performed by everyone except for the seriously disabled or very frail. Smartphones and their embedded computer technologies are increasingly being used to promote physical activity. Gamification presents itself as a promising approach to overcome a loss of interest, increase user engagement , raise the quality of health behaviors , and motivate users to use mHealth apps for a sustained period

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria were 18 to less than 60 years of age,
* under- going conventional hemodialysis three times a week,
* hemodialysis period of three month or more,
* having smartphone aneroid access (second group),
* Available for telephone follow-up ,
* ability to read and write ,
* and being ambulatory,
* Patients using a cane or other assistive device will be eligible and Patients provided informed consent to participate.

Exclusion Criteria:

The study will exclude patients with

* unstable angina,
* those with lower-limb amputation
* and those using wheelchairs.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 94 (Actual)
Dates: Start 2022-10-31 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
change in patients weekly step count | will be measured at baseline and after intervention [(after 12 weeks of walking program)]
  Step count will be assessed using a pedometer.
change in fatigue level | will be measured at baseline and after intervention [(after 12 weeks of walking program)]
  Brief Fatigue Inventory questionnaire will evaluate the level of current fatigue and usual fatigue in the last 24 hours.A score of 0 means no fatigue and a score of 10 means the highest level of fatigue. The total score of fatigue was obtained through summing up the score of questions 2e10 (nine items) and dividing by nine

SECONDARY OUTCOMES:
change in sleep quality | will be measured at baseline and after intervention [(after 12 weeks of walking program)]
  Sleep disorders will be assessed using the arabic version of the Pittsburgh Sleep Quality index (PSQI).The scores were added to yield a global PSQI score in the range 0-21, with a higher score indicating poorer sleep quality.
change in functional status | will be measured at baseline and after intervention [(after 12 weeks of walking program)]
  The Short Physical Performance Battery (SPPB) is designed to measure functional status and physical performance.Each task is scored out of 4, with the scores from the three tests summed to give a total, with a maximum of 12 and a minimum of 0. A higher score indicates a higher level of function, while lower scores indicate a lower level of function
change in heart rate | will be measured at baseline and after intervention [(after 12 weeks of walking program)]
  a checklist to assess heart rate
change in respiratory rate | will be measured at baseline and after intervention [(after 12 weeks of walking program)]
  a checklist to assess respiratory rate
change in systolic blood pressure | will be measured at baseline and after intervention [(after 12 weeks of walking program)]
  a checklist to assess systolic blood pressure
change in diastolic blood pressure | will be measured at baseline and after intervention [(after 12 weeks of walking program)]
  a checklist to assess diastolic blood pressure

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Nursing Mansoura University, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Elzeky MEH, Ramadan El-Shaboury RH, Salameh B, Samaan E, F M Shahine N, Abdelhamid A. Effects of gamified versus pedometer-based walking intervention on physical activity, fatigue, and sleep quality among hemodialysis patients: a quasi-experimental study. BMC Nephrol. 2025 Mar 3;26(1):108. doi: 10.1186/s12882-025-04012-7. PMID 40033223